CLINICAL TRIAL: NCT01116245
Title: A Randomized, Single Blind, Placebo Controlled Phase 2 Study to Assess the Safety of ADXS11-001 for the Treatment of Cervical Intraepithelial Neoplasia Grade 2/3
Brief Title: An Assessment of an Attenuated Live Listeria Vaccine in CIN 2+
Acronym: ADXS11-001
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to lack of enrollment
Sponsor: Advaxis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lm-LLO-E7-07
Record Dates: First submitted 2010-04-20; First posted 2010-05-04 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervical Intraepithelial Neoplasia Stage 2/3
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low Dose (Experimental): 5x10^7 cfu x 3 intravenous infusions at 28 day intervals. All infusions will be preceded by prophylactic NSAID and antihistamine, and followed 3d later with antibiotic.
  Interventions: Biological: ADXS11-001 (Lm-LLO-E7)
- Middle Dose (Experimental): 3.3x10^8 cfu x 3 intravenous infusions at 28 day intervals. All infusions will be preceded by prophylactic NSAID and antihistamine, and followed 3d later with antibiotic.
  Interventions: Biological: ADXS11-001 (Lm-LLO-E7)
- High Dose (Experimental): 1x10^9 cfu x 3 intravenous infusions at 28 day intervals. All infusions will be preceded by prophylactic NSAID and antihistamine, and followed 3d later with antibiotic.
  Interventions: Biological: ADXS11-001 (Lm-LLO-E7)
- Placebo (Placebo Comparator): normal saline x 3 intravenous infusions at 28 day intervals. All infusions will be preceded by prophylactic NSAID and antihistamine, and followed 3d later with antibiotic.
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Biological: ADXS11-001 (Lm-LLO-E7) — ADXS11-001 at one of three dose levels given as 3 vaccinations separated by 4 weeks with an oral antibiotic regimen subsequent to dosing.
  Arms: High Dose; Low Dose; Middle Dose
Drug: Placebo Control — 3 intravenous infusions of normal saline at 28 day intervals. All infusions will be preceded by prophylactic NSAID and antihistamine, and followed 3d later with antibiotic.
  Arms: Placebo

SUMMARY:
Cervical cancer is associated with Human Papilloma Virus. About 57% of cervical cancer is the result of infection by Human Papilloma Virus strain 16 (HPV-16). HPV is a very common virus that can affect the cells of the cervix. E7 is a substance that is made by the HPV virus which causes cervical cancer. The purpose of the study is to test the safety, tolerability (how the drug makes you feel), immunology (effects on the immune system) and efficacy (disease curing effects) of a vaccine called Lovaxin C against E7. The vaccine is designed to cause the immune system to react against the E7 substance in a manner that is intended to reverse the changes to the cervix and prevent cervical cancer from occurring.

DETAILED DESCRIPTION:
Worldwide, many women carry HPV and cervical cancer is the leading cancer killer of women under the age of 50. Although its consequences are considerably less severe in the US, it leads to considerable morbidity. Many published clinical trials describe the immunotherapeutic treatment of early stage, pre-invasive, cervical cancer. It is widely recognized that immunotherapies are most effective in early stage disease because the immune system is least debilitated and disease burden is lowest. Invasive cervical cancer is preceded by a long, slowly progressive, pre-invasive phase termed Cervical Intraepithelial Neoplasia (CIN), which allows for this therapeutic approach. An ideal therapy would result in the remission of CIN 2/3 without damage to cervical tissue. A National Institute of Cancer panel charged with achieving consensus on this issue concluded that a non-surgical medical treatment for this indication would be valuable

The primary objectives of this trial are to test three doses of Lovaxin C to determine if vaccination with Lovaxin C in women with CIN 2/3 for whom surgery is indicated can safely reverse the disease compared to placebo treated control patients.

An earlier Phase 1/2 trial of Lovaxin-C in late stage metastatic cervical cancer used a regimen of two doses given with a 28-day interval. That regimen was shown to be safe and to generate reduction in tumor burdens in some patients. In this trial we will treat earlier stage disease in healthier patients with better immune systems, will use the same and lower doses as given before, but add an additional dosing to the regimen by administering the lowest dose that we assessed previously and by adding a third vaccination to the prior regimen. Unlike the phase 1 trial in which 2 doses were given with a 3 week separation, dosing in the proposed trial will be separated by 4-week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CIN 2/3 that requires surgical intervention

Exclusion Criteria:

* Previous history of listeriosis
* Steroid use
* Antibiotic use
* Negative anergy panel
* HIV positive
* Pregnant or actively trying during the treatment period
* Intercurrent disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The primary end point will be a histologic determination of whether CIN 2/3 present at entry had regressed. | 11 months

SECONDARY OUTCOMES:
Secondary efficacy endpoints include whether HPV DNA was reduced or eliminated and a comparison of their excised cervical tissue controls to assess the extent of disease in treated vs. untreated patients. | 11 months

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - New Horizons Women's Care, LLC, Chandler, Arizona
  - Arizona OB/GYN Affiliates, PC, Phoenix, Arizona
  - Precision Trials, Phoenix, Arizona
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Grossmont Center for Clinical Research, La Mesa, California
  - Visions Clinical Research, Boynton Beach, Florida
  - Altus Research, Lake Worth, Florida
  - Center for Women, Chicago, Illinois
  - Indiana University Dept. of OB/GYN Oncology, Indianapolis, Indiana
  - New York Downtown Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Temple University, Philadelphia, Pennsylvania
  - InVisions Consultants, LLC- c/o Institute for Women's Health, San Antonio, Texas
  - InVisions Consultants, LLC, San Antonio, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah